CLINICAL TRIAL: NCT01166048
Title: Randomized Double-blind Study Comparing the Efficacy of Duloxetine With Placebo in Patients With Chronic Low Back Pain With a Radicular Component
Brief Title: Comparison of the Efficacy of Duloxetine With Placebo in Patients With Chronic Low Back Pain With a Radicular Component
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sibylle Pramhas, MD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPDP-01
Record Dates: First submitted 2010-05-18; First posted 2010-07-20 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Radicular component; neuropathic pain; duloxetine; CLBP
MeSH Terms: conditions — Neuralgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milk powder pill (Placebo Comparator): Patients will receive 2 placebo pills per day for a period of 4 weeks.
  Interventions: Drug: Duloxetine
- Duloxetine (Experimental): In the experimental arm of the study patients will receive duloxetine, which will be titrated up to a dosage of 120mg over a period of two weeks and continued at this dosage for two weeks.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Patients will receive 120mg of Duloxetine for the duration of 2 weeks after a dosage titration of 2 weeks according to the following scheme: (p=placebo)
  day: 1 2 3 4 5 6 7: p-30mg p-30mg p-30mg p-30 mg p-30mg p-30mg p-60mg
  day: 8 9 10 11 12 13 14: p-60 mg p-60 mg p-60mg p-60mg p-60mg p-60mg 60-60mg
  Arms: Milk powder pill
Drug: Duloxetine — 2 weeks of titration of duloxetine to 120mg, (1-0-1), 2 weeks of continuation on 120mg/day.

SUMMARY:
Objective:

The objective of this study is to compare the efficacy of duloxetine in the treatment of patients with chronic low back pain with a radicular component to placebo.

Study hypothesis:

Duloxetine is a new substance now in use for the treatment of neuropathic pain. It has proven its efficacy in diabetic peripheral neuropathy and fibromyalgia in several trials. The investigators therefore hypothesize that duloxetine will be efficacious in patients with chronic low back pain and a radicular component.

Study Rationale:

Chronic low back pain is an extremely common diagnosis. However, therapeutic options for the condition are limited and therapy remains difficult. Duloxetine has proven its efficacy in patients with neuropathic pain and may also be useful in chronic low back pain. If the investigators are able to show a benefit for patients in the duloxetine arm, the substance may constitute a further treatment alternative in chronic low back pain.

Study Design:

Prospective, randomized, double-blind placebo-controlled cross over study. Patients will be administered duloxetine for 4 weeks followed by a 2 week wash-out phase after which they will be medicated with placebo for 4 weeks. A second group of patients will receive the medication in reversed order. The primary study endpoint is constituted the weekly mean of VAS-Score in the last week of each treatment period. Secondary endpoints are defined as use of rescue medication, Beck Depression Inventory score, Health related Quality of Life SF-36 score and side effects/adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ( below L1)
* Chronic pain, >6 months
* Visual Analogue Scale (VAS) ≥ 5
* Back pain with radicular component defined as pain with a burning, tingling sensation within the anatomic distribution of the nerve root and diagnosed by painDETECT questionnaire
* Failed back surgery

Exclusion Criteria:

* Current mood disorder (dysthymia, bipolar mood disorder)
* Major Depression > 12 months (Beck Depression Inventory Score ≥ 18)
* History of a psychoactive substance use disorder within the preceding 12 months
* Major coexisting medical illness (e.g. severe heart failure, pulmonary hypertension, renal insufficiency)
* Glaucoma
* Acute myocardial infarction
* uncontrolled hypertension
* Prostate hyperplasia
* History of convulsion
* Pregnancy; women of childbearing age will be required to use contraceptives during the duration of the study. Furthermore a pregnancy test will be performed prior to the beginning of the study and once a month during the study period.
* Participation in a clinical trial in the 3 weeks preceding the study
* Allergy to study medication
* Use of the following medication:

  * opioids except for tramadol,
  * benzodiazepines other than indicated at low doses for sleep disorders
  * antineuropathic medication including except for that specified in the study protocol
  * muscle relaxants
  * antidepressants other than indicated at low doses for sleep disorders
  * NSAID, Paracetamol
  * non-selective MAO-Inhibitors
  * Fluvoxamine, Ciprofloxacin, Enoxacin
  * Selective Serotonin-reuptake Inhibitors (SSRI)

if tapering of these drugs is impossible before inclusion.

* Impaired kidney function (Creatinine > 1.5mg/dl)
* Impaired hepatic function (GOT, GPT >2 fold standard levels)
* Patients who are not able to understand the study measures and are not able to complete pain assessment forms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Weekly mean pain intensity in study phase I (Visual analogue score, units 1-10) | Week 4 of study period
  Operationally a VAS is a horizontal line, 100 mm in length, anchored by word descriptors at each end (left= no pain, right=worst imaginable pain).The patient marks the current subjective pain intensity on the scale. This is converted to a numeric value by measurement from the left side of the scale. (Units 1-10)
Weekly mean pain intensity in study phase II (Visual analogue score, units 1-10) | Week 10 of study period

SECONDARY OUTCOMES:
Use of rescue medication in study phase I | Use of rescue medication in week 4 of study period
  Patients will be allowed Metamizol (500mg up to 3g per day) and Tramadol drops (20 ggt. up to 6 times per day) as rescue medication. Rescue medication will be recorded daily in a patient diary. Use of rescue medication will be scored as follows: 0=no rescue medication; 1=metamizol; 2=tramadol
Beck Depression Inventory score in phase I of study period | Beck Depression Inventory score at week 4 of study period
  Subjects will be asked to perform the Beck Depression Inventory at screening and at week 4.
Health related Quality of Life SF-36 score in phase I of study period | Health related Quality of Life SF-36 score at week 4 of study period.
  Subjects will be asked to fill out the Health related Quality of Life SF-36 questionnaire at screening and at the end of each treatment period (placebo and verum)
painDetect score in phase I of study period | painDetect score at week 4 of study period.
  Subjects will be asked to complete the painDetect questionnaire at screening and the end of each treatment period (placebo and verum).
Use of rescue medication in phase II of study period | Use of rescue medication in week 10 of study period.
Beck Depression Inventory score in phase II of study period | Beck Depression Inventory score at week 10 of study period.
Health related Quality of Life SF-36 score in phase II of study period. | Health related Quality of Life SF-36 score at week 10 of study period.
painDetect score in phase II of study period | painDetect score at week 10 of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Oehmke, MD, Principal Investigator — Department of Special Anesthesia and Pain Therapy, Medical University of Vienna, AKH Vienna,
Locations (1):
- Department of Special Anesthesia and Pain Therapy, Medical University of Vienna, AKH Vienna, Vienna, Vienna, Austria